CLINICAL TRIAL: NCT04132778
Title: A Novel Digital Self-management System Targeting Automated Prevention of Asthma
Brief Title: Digital Prevention of Asthma
Acronym: AsthmaTuner
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The recruitment stopped due insufficient funding.
Sponsor: Karolinska Institutet (Other)
Collaborators: Tiohundra AB (Industry); Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Björn Nordlund, Research group leader, co-founder of the investigational product, PhD and RN, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: v.10
Record Dates: First submitted 2019-10-14; First posted 2019-10-21 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2023-02

CONDITIONS: Asthma; Care Management, Patient
Keywords: Asthma; AsthmaTuner; Management
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: RCT with two arms, Asthmatuner or traditional asthma management, during at least 6 months. Thereafter, the study continues to be observational from 6- 12 months.
Who Masked: Investigator
Masking Description: Physician blinded to the allcocated treatment; AsthmaTuner or traditional treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention - Asthmatuner (Experimental): Asthmatuner (Medituner AB, Stockholm, Sweden) is a CE-marked cloud-computing-based system with a healthcare interface and a downloadable patient app (Android or iOS).The intended use of Asthmatuner is to automate asthma self-management by letting patients register symptoms and measure forced expiratory volume in one second (FEV1) with a Bluetooth spirometer (MIR, SmartOne). The patient then receives immediate feedback on the status of symptom control (controlled, partly controlled or uncontrolled), and a treatment recommendation, with an image of the correct inhaler or other type of medication and the dose. Symptom control is quantified based on lung function; litre to percentage of personalised best FEV1, using a cut-off ≤80% and symptoms during the last week based on four questions: 1) need for rescue medication more than twice due to asthma symptoms, 2) any daytime symptoms, 3) nocturnal symptoms/awakenings, and 4) limitation in physical activities.
  Interventions: Device: AsthmaTuner
- Control group - Traditional asthma management (No Intervention): Traditional self-management is defined as all other types of non-digital asthma management. This could be treatment plan written on paper or by oral communication to patient/caregiver on asthma treatment.

INTERVENTIONS:
Device: AsthmaTuner — Conventional treatment was defined as non-digital self-management using paper individual treatment plans, which contained treatment adjustments of prescribed medications according to symptoms of controlled, partly controlled or uncontrolled asthma, along with instructions according to national guidelines.
  Other Names: Digital Automated self-management
  Arms: Intervention - Asthmatuner

SUMMARY:
Asthma self-management is dependent on support and education. To facilitate self-management have we developed and CE-mark a novel digital self-management system called Asthmatuner (Medituner AB, Sweden).The primary aim of this program is to evaluate if self-management with Asthmatuner improves asthma control more than traditional self-management. RCT with two arms, Asthmatuner or traditional asthma management, during at least 6 months. Thereafter, the study continues to be observational from 6- 12 months. Eligible patients with doctor's diagnosed asthma that are managed within the municipality of Tiohundra and Astrid Lindgren Children's Hospital will be invited to participate. Approximately 800 patients, adults and schoolchildren of the age of 6 years will be recruited.Outcomes: Asthma Control Test, number of exacerbations, unplanned healthcare visits, Medicine Adherence Report Scale and lung function.

DETAILED DESCRIPTION:
The ultimate goal for all patients is to achieve asthma control. There are various tools for evaluating a patient's asthma control, one is to use validated questionnaires e.g. Asthma Control Test (ACT) (1), another is to evaluate symptoms in patient history based on recommended characteristics from the Global Initiative for Asthma (GINA) (2). These characteristics emphasize optimal asthma control as no symptoms, undisturbed sleep, no severe exacerbations, no emergency visits, normal lung function and no limitations in daily activities.

The characteristics defining asthma control according to GINA guidelines are widely used as the golden standard for both clinical research and for asthma care (3, 4). Based on a patient's number of characteristics, GINA classifies asthma as controlled, partly controlled or uncontrolled (5). The GINA guidelines include two domains for assessment, the first is the evaluation of symptoms and the second is physician´s evaluation of patient's future risk for exacerbations. Indicators of increased health cost of asthma like e.g. health care utilization, medication and lost school/work days are associated with uncontrolled asthma (6). In addition, studies have shown that patients with lower socio-economic status are associated with more impaired asthma control (7-9), and further attention is needed to assist patients with impaired asthma control through new approaches and better management strategies.

Poor adherence to asthma management and simple practical tools for diagnosing asthma can lead to under- and over-diagnosis of asthma in primary health care (10, 11). In most cases, including in the EU, asthma patients visit their doctors less than once a year, giving healthcare providers only a snapshot of the patient's condition (12, 13). New approaches are needed to improve adherence in asthma care.

Patient education in self-management using self-monitoring of lung function and symptoms, coupled with adjustable treatment plan appear to be effective compared with other forms of asthma self-management according to a Cochrane review (14). National asthma programmes focusing on management and improving asthma care has proved to reduce the morbidity of asthma and its impact on individuals as well as on the society (15). Patient education in self-management improves health and the quality of life for people with asthma, as well as reducing health care costs (14). However, in spite of this convincing evidence on how to treat and manage asthma, there is worldwide significant discrepancy between real life practice and guidelines of asthma management (16, 17).

Clinical decision support systems for self-management Significant worldwide discrepancy exists between real life asthma practice and guidelines of management (16, 17). Self-management based on self-monitoring of lung function and symptoms, coupled with adjustable treatment plan appear to be effective compared with other forms of asthma self-management according to a Cochrane review (14). Furthermore, electronic medical records are largely implemented in asthma care, and it is feasible to enable health care providers to monitor and support patient's self-management with computer decision support systems (CDSS). Therefore, we target to improve incomplete asthma management by develop and CE-mark the novel digital self-management system Asthmatuner (Medituner AB, Sweden). The system consists of a patient smartphone application and a portable wireless spirometer for measuring lung function, and a healthcare provider user interface to prescribe treatment plan and assess patient data. The app provides patients with a daily treatment recommendation linked to patient's current status of asthma (controlled, partly- or uncontrolled asthma) (2). Recently in 2018, Asthmatuner significantly reduced asthma symptoms in children and adolescents compared to traditional management in a randomised controlled cross-over trial (18).

Prevention of exacerbations and symptoms is major health care challenge. Combining data from a variety of sources, including risk factors and real-time biological and environmental data has the potential to improve the prediction of asthma attacks in individuals. Quantifying time-serial measures of lung function contain unexpected amounts of information that can be linked to occurrence of symptoms and exacerbations (19). Thus, our hypothesis is that Asthmatuner constitutes a unique data source that offers identification of longitudinal fluctuating patterns of lung function that can be used to develop algorithms capable of predicting airway obstruction and generating early individual-specific action plan. Individual action plan could contain phenotype specific information about step-up treatment, reminders on how to use and inhaler medication and avoiding specific factors that may trigger or worsen asthma symptoms, as well as contact details for healthcare providers (20). In addition, Asthmatuner has the potential to strengthen quality in primary health care at reduced cost (21), by identify patients with poor asthma control and therefore most needed for clinical follow-up or video online visit. Therefore, the municipality of Tiohundra (22), with a population of more 56000 people, has decided to assess the effect and benefit of using Asthmatuner in a randomised controlled trial (RCT).

The primary aim of this program is to evaluate if self-management with Asthmatuner improves asthma control more than traditional self-management.

Secondary aims are to:

* Evaluate if Asthmatuner can reduce the number of planned or unplanned health care visits compared with traditional asthma care
* Investigate if Asthmatuner improves adherence to intake of control medication and health-related quality of life (HR-QoL) more than traditional traditional asthma care
* Assess if Asthmatuner can reduced the number of exacerbations and missed work/school days due to asthma compared with traditional asthma care
* Characterise specific phenotypes based on biodata and time-serial measurements of lung function in relation to occurrence of symptoms and exacerbation in patients using Asthmatuner. The goal is to develop mathematical algorithms generating action plan for prevention of exacerbation. Moreover, the data collected with Asthmatuner and the daily treatment recommendations generated with this system will be used to train a deep (artificial) neural network towards an optimization of the ACT scores (i.e., the level of asthma control) attained.
* Perform a qualitative study with the third and final aim to explore patients' and caregivers' experience of using Asthmatuner

MATERIAL AND METHODS Design RCT with two arms, Asthmatuner or traditional asthma management, during at least 6 months. Thereafter, the study continues to be observational from 6- 12 months, offering all willing participants to use Asthmatuner. In addition, a complementary qualitative study of patients' and caregivers' experiences of the introduction and use of Asthmatuner and its impact on work processes and communication.

Primary outcomes at baseline, 3- and 6 months study period

* Mean score validated Asthma Control Test (ACT) Secondary outcomes by 6 months study period
* Number of exacerbations requiring oral corticosteroids or health care utilisation
* Unplanned health care visits due to asthma
* Mean score of Mini-Asthma Quality of Life Questionnaire (Mini-AQLQ)
* Mean score of Medicine Adherence Report Scale
* Fluctuation in time-serial measurements (forced expiratory volume in one second FEV1 (L)) with use of Asthmatuner, linked to information about exacerbations and daily or nocturnal symptoms or treatment with bronchodilator
* Cost benefit with Asthmatuner compared with traditional health care visits based on costs for planned/unplanned visits, exacerbations, and effect on ACT
* Patient and caregiver satisfaction with Asthmatuner. using survey and interviews after completed study participation.

The qualitative study will focus on patients' experiences (eg patient satisfaction, empowerment, communication with healthcare professionals and perceived quality of care) as well as the caregivers' experiences (eg work processes, perceived stress, impact on communication and perceived quality of care).

Subjects Primary care Eligible patients with doctor's diagnosed asthma that are managed at any health care centre within the municipality of Tiohundra will be invited to participate. Approximately 400 patients, adults and schoolchildren of the age of 6 years will be included. Subjects with untreated or treated comorbidity with major effect on the state of asthma will not be included.

Paediatric cohort The study population will be extended to 400 schoolchildren with asthma to ensuring sufficient number of participants and time-serial measurements of lung function. Children and adolescents 6-18 years, at Astrid Lindgren Children's Hospital in Stockholm (Karolinska University Hospital) will be invited to attend during the year 2019-2020.

Sample Size The sample size for the trial will be estimated based on our pilot study showing that Asthmatuner improves asthma control with 3.72 ACT points compared to traditional management 2.35 points (mean standard deviation 3.45). Assuming a dropout rate up to 10%, including 200 eligible subjects for Asthmatuner and equal number in the control group would be clinical relevant, worthwhile and feasible to attain 80% power at 5% significant level.

Intervention - Asthmatuner Patients download the app from AppStore or Google Play and create a user account. The healthcare provider must also have access to patients' Asthmatuner accounts so the doctor or asthma nurse can ensure the treatment plan is up to date. The patient will then be able to see the treatment plan and which inhaler they should use displayed on the screen of the smartphone. The smartphone application has been designed to minimize the time needed to generate an individual treatment recommendation. Once the user profile has been created, the wireless spirometer is paired with the smartphone and the physician creates and uploads a treatment plan based on an automated recommendation, which is generated in seconds.

The user interface is intuitively structured into four sections: 1) Lung function, 2) Symptoms, 3) Treatment, and 4) Trends view.

To get an up-to-date treatment recommendation the patient follows the instructions on the screen under the Lung function section to generate an FEV1 (Forced Expiratory Volume) value using the connected spirometer from MIR (Medical International Research, Italy). The interface shows if the value was correctly generated and how it relates to patient's personal best value. Four symptom questions - in accordance with the GINA - are presented and the patient answers yes or no. Once the symptom questions have been saved, the patient is automatically transferred to the "treatment section" where the current treatment recommendation is presented based on lung function and symptoms. The trend feature shows the patient/provider a historical overview of lung function, symptoms and treatment.

Control group - Traditional asthma management Traditional self-management is defined as all other types of non-digital asthma management. This could be treatment plan written on paper or by oral communication to patient/caregiver on asthma treatment.

Registers Complementary information about unplanned visits and health care utilisation both in-patient care and out-patient care in Sweden will be collected from the medical record Take Care or the National Quality Register for Asthma and COPD "Luftvägsregistret". The study will be registered at ClinicalTrials.gov.

Asthma control test Asthma symptoms during the last 4 weeks will be assessed using Childhood asthma control test (C-ACT) in children 6-11 years and ACT patients aged > 12 years. The questionnaire is validated and regular used in clinical practice (23). Well-controlled asthma is defined as score > 20 points and uncontrolled asthma score of < 19.

Health survey Health survey including socio-demographics, medical history about asthma, comorbidities and symptoms, as well as ACT will be filled out by patient/caregiver at inclusion.

Electronic questionnaires Questionnaires will be sent out electronically by use of KI-survey, collecting information on ACT, symptoms, exacerbations, unplanned health care visits/consultations due asthma, loss of work and school days due to asthma at 3 and 6 months.

Health-related quality of life (HR-QoL) HR-QoL will be applied at baseline, 3- and 6 months using the validated Swedish translated the Mini-AQLQ in patients from 12 years of age (24).

The MARS questionnaire Self-reported medication adherence will be measured with validated five-item MARS, developed to assess adherence with asthma medication (25). The MARS comprises statements about medication use behaviors. The patient is asked to answer each behavior with a score between 1-5 based on of following alternatives; "always", "often", "sometimes", "rarely" or "never". A mean MARS score will then be calculated, and a score of 4.5 or greater indicates good adherence (25).

Lung function testing Lung function will be measured at each study visit, analysing FEV1, forced vital capacity (FVC), FEV1/FVC and forced expiratory flow after 25-75% of vital capacity (FEF25-75). At visit 1 is a reversibility test performed after intake short-acting beta-2 agonist.

Follow-up visits Frequency of follow-up visits and management are recommended according to Swedish National Board of Health and Welfare, Table 3.

Statistical analysis Statistical analysis will be carried out analysing proportion of subjects maintaining asthma control or improving their asthma control according to ACT and GINA between management groups, as well as the numeric change in ACT scores from baseline to study end.

Methods of computational methodology

The fluctuation-based clustering (FBC) method consists of identifying clusters of patients with similar patterns of lung function fluctuation by comparing each patient's empirical distribution of daily lung function measurements recorded over a predetermined window of observation. The FBC method has been described in detail elsewhere (26). In brief, this approach consists of the following steps:

1. Quantification of similarity in lung function fluctuation between individuals; and
2. Grouping of individuals into clusters such that similarity between members of the same cluster is strong and between different clusters is weak.

Furthermore, the FBC method includes a data-driven process for determining the tolerable amount of missing measurements. It starts with the selection of a highly compliant subset of patients (i.e. with a high number of performed lung function measurements, normally with at least as many measurements as the 60th percentile of the overall distribution of the number of lung function measurements from the entire analysis population), the so-called gold standard. Then, within the gold standard, to quantify similarities in lung function fluctuation between individuals, the distribution of normalised lung function values of a given patient is compared with the distributions of all other patients in the gold standard. This pairwise comparison is done using the earth mover's distance. A low value of earth mover's distance indicates high similarity in lung function fluctuation between two individuals. Patients are then grouped into clusters, such that the similarity between members of the same clusters is strong while that between different clusters is weak, using Ward's minimum-variance hierarchical clustering method. Following this, a cluster stability analysis is performed to assess the stability of the clusters upon random data point removal. The outcome of this stability analysis enables us to establish the minimum number of lung function measurements required to ensure the clusters' stability. Those patients who performed the minimum number of lung function measurements required but were not part of the gold standard are now added to the gold standard. Finally, the cluster analysis procedure is repeated with this extended gold standard to obtain the final clusters.

Monitoring plan Before the beginning of the investigation, the Sponsor will appoint an independent monitor. Monitoring will be performed before, during the study and after the study is completed in accordance with the ISO 141 55 GCP (Good Clinical Practice) standard. Study conductance, source data, device accountability, adherence to the study protocol, Good Clinical Practice, and regulatory requirements will be monitored in approximately 30-50% of all included subjects.

Data to be monitored at site are e.g.

* Patient information and Informed Consent. That patient included in the study has signed an Informed Consent and that no study procedures have begun before the date of the consent.
* That inclusion and exclusion criteria are met for the included patients that are monitored
* That all types of adverse events and serious adverse events, device related or not, as well as, those that might have led to SAE shall be reported.
* Check that CRF data are entered in those subjects that are monitored
* Other CRF data will be source data verified against patient records according to a detailed Monitoring Plan (that will contain details regarding the overall monitoring) signed by the Sponsor prior to the start of the study. At least 20% of the patients will have data in the CRFs 100% source data verified.

The monitor and possible authorities must be given direct access to source documents (original documents, data and records). Direct access includes permission to examine, analyse, verify and reproduce any record(s) and report(s) that are important to the evaluation of the clinical investigation. In order to be able to do that, a written consent from each patient should be obtained. Also a secrecy agreement between the monitor and the person responsible for patient records at the study site will be signed.

Data management Procedures for data management will be implemented in collaboration with KTA and conducted according to standards of GCP. Due to work load and the nature of the intervention, neither health care personnel nor participants can be blinded to allocation. An employee outside the research team will feed data into the computer in separate datasheets so that the researchers can analyse data without having access to information about the allocation.

Database cleaning and issuing data queries will be traceable and transparent with logs and data is stored at Karolinska Institutet, department of Women's and Children's Health. Audit will be performed once by certified CRO to assure quality, and to verify the monitoring process and data as appropriate.

Paper case report forms (CRF) will be completed for each included patient in combination with standardized health questionnaires at baseline, together with validated ACT at 3- and 6 or later after study inclusion. Investigators will ensure completion and review of the CRF. Investigators have personal responsibility for the accuracy and authenticity of all clinical and other data that are entered into the CRF. Subjects included in the study will be desidentified on the CRFs and subsequent reporting. A Subject Identification List, with cross reference between the subjects identification number in the study and the subjects personal data, will be kept looked away with the study documentation at the study centre. Monitors will do on site monitoring to review the data in the CRFs versus source data and issue queries to the Investigator to correct and clean data before CRF is sent to be entered into the a database, stored and kept by the Sponsor. The study database will be reviewed and cleaned prior to locking the study database and analysing the data, and a Clean File Report will be issued. During the course of the study the investigational team, and the monitor will have access to the study material, which will be kept in a locked place. Retention period for data storage is 10 years. All study documentation will be saved as paper copies and electronic files after the study has been published and reported. Participating investigators / Sponsor will be responsible for data collection, data processing and report writing.

Adverse events, adverse device effect and device deficiencies

DEFINITIONS of categories of adverse events from ISO/FDIS 14155:

Adverse Device Effect (ADE) is an adverse event related to the use of Asthmatuner:

NOTE 1- This includes any adverse event resulting from insufficiencies or inadequacies in the instructions for use, the deployment, the implantation, the installation, the operation, or any malfunction of the investigational medical device.

NOTE 2- This includes any event that is a result of a use error or intentional misuse.

Adverse Event (AE) is any untoward medical occurrence, unintended disease or injury or any untoward clinical signs (including an abnormal laboratory finding) in subjects, users or other persons whether or not related to the investigational medical device:

NOTE 1: This includes events related to the investigational device or the comparator.

NOTE 2: This includes events related to the procedures involved (any procedure in the clinical investigation plan).

NOTE 3: For users or other persons this is restricted to events related to the investigational medical device.

Device deficiency is inadequacy of a medical device related to its identity, quality, durability, reliability, safety or performance, such as malfunction, misuse or use error and inadequate labeling. Investigational medical device Asthmatuner will in this clinical investigation be assessed for safety or performance.

Serious Adverse Device Effect (SADE) is adverse device effect that has resulted in any of the consequences characteristic of a serious adverse event.

Serious Adverse Event (SAE) is an adverse event that:

1. led to a death,
2. led to a serious deterioration in health that either:

   1. resulted in a life-threatening illness or injury, or
   2. resulted in a permanent impairment of a body structure or a body function, or
   3. required in-patient hospitalization or prolongation of existing hospitalization, or
   4. resulted in medical or surgical intervention to prevent life threatening illness or injury or permanent impairment to a body structure or a body function.
3. led to fetal distress, fetal death or a congenital abnormality or birth defect.

NOTE 1: This includes device deficiencies that might have led to a serious adverse event if a) suitable action had not been taken or b) intervention had not been made or c) if circumstances had been less fortunate. These are handled under the SAE reporting system.

NOTE 2: A planned hospitalization for pre-existing condition, or a procedure required by the Clinical Investigation Plan, without a serious deterioration in health, is not considered to be a serious adverse event.

Unanticipated Serious Adverse Device Effect is serious adverse device effect which by its nature, incidence, severity or outcome has not been identified in the current version of the risk analysis report.

NOTE: Anticipated: an effect which by its nature, incidence, severity or outcome has been previously identified in the risk analysis report

Reportable events according 90/385/EEC and 93/42EEC. The following events are considered reportable events based on definitions above:

* any SAE
* any Device Defieciency that might have led to a SAE if a) suitable action had not been taken or b) intervention had not been made or c) if circumstances had been less fortunate
* new findings/updates in relation to already reported events

Report by whom: Reportable events have to be reported by the sponsor of the clinical investigation, which could be the manufacturer, the authorized representative or another person or entity.

Report to whom: Reportable events must be reported at the same time to all NCA where the clinical investigation has commenced using the summary tabulation featured in the Appendix 4. A list of clinical investigation contact points within the NCA's is published at the Commission's homepage (http://ec.europa.eu/growth/sectors/medical-devices/contacts/index_en.htm), access date: 2016-02-22

Reporting timelines

The sponsor must report to the NCAs where the clinical investigation has commenced:

* a SAE which indicates an imminent risk of death, serious injury, or serious illness and that requires prompt remedial action for other patients/subjects, users or other persons or a new finding to is: immediately, but not later than 2 calender days after awareness by sponsor of a new reportable event or of new information in relation with an already reported event.
* any other reportable events as described in section "Reportable events according 90/385/EEC and 93/42EEC" or a new finiding/update to it: immediately, but not later than 7 calendar days following the date of awareness by the sponsor of new reportable event or of new information in relation with an already reported event.

Report by the investigator to the sponsor The sponsor will implement and maintain a system consisting of email address and phone number to sponsor, to ensure that the reporting of the reportable events will be provided by the investigator to the sponsor in acceptable timely conditions, but not later than within 3 calendar days after the occurrence of the event.

Reporting form The reporting form template for the summary SAE tabulation is given in the Appendix 4 of this document. The table gives a cumulative overview of the reportable events per clinical investigation and will be updated and transmitted to participating NCAs each time a new reportable event or a new finding to an already reported event is to be reported. More detailed information has to be provided on request of an NCA.

The sponsor shall identify the new/updated information in the status column of the tabular form featured in the Appendix 4 as:

a = added = new reportable event; m = modified = new finding/update to an already reported event; u = unchanged. Changes in a line should be highlighted in bold and/or color in the respective column. English is the recommended language for the reporting form. The report should be sent by email.

Preexisting conditions and unanticipated adverse device effects In this trial, a preexisting condition i.e. asthma, should not be reported as an adverse event unless the condition worsens or episodes increases (i.e. exacerbations) in the frequency during the adverse event reporting period.

Procedures Diagnostics and therapeutic non-invasive and invasive procedures, such as surgery, should not be reported as adverse events. However, the medical condition for which the procedure was performed should be reported if it meets the definition of an AE. The AE reporting period begins upon starting the use of Asthmatuner or conventional management (visit 1).

Each participant will be questioned about AE for each visit. All AE that occur in the trial should be reported to investigator and specified in the participants´ medical journal and in a separate AE form with following information:

* Type of AE
* Date and time of AE
* Association with Asthmatuner (No/Yes/Unknown)
* Gravity (Serious or Non-serious)
* Reporting time
* Follow-up (resolved or unresolved)

Contact details for reporting serious AE:

1. Björn Nordlund, RN and PhD, Department for Women's and Children's Health, Karolinska Institutet. Phone: +46 703234414
2. Henrik Ljungberg, MD and PhD, Astrid Lindgren Children's Hospital, Lung-Allergy Department and Department for Women's and Children's Health, Karolinska Institutet. Phone: +46 706628642 QUALITATIVE STUDY - PROCEDURES Before the introduction of Asthmatuner, caregivers will be interviewed focusing on their expectations. After at least 6 months, caregivers and patients will be interviewed with regard to how they experienced the use of Asthmatuner. All caregivers within Tiohundra's primary care that work with asthma/COPD patients are asked about participation in the interview study. The patient selection for the qualitative part is done among adult patients with asthma diagnosis who are randomized to use Asthmatuner. They will have mixed disease history, sex and age for maximum selection width.

For participation in the qualitative study, the participants will be informed that all participation is voluntary and can be discontinued when and without any specific reason. The participants who are patients will be asked at the primary care center in connection with the planned visit, or be contacted via letter for participation in the interview. The responsible doctor, nurse or researcher obtains informed written consent after the research subjects have received sufficient time for consideration. When the caregivers are informed about the study, participation in the qualitative study is offered. Information is then given that all participation is voluntary and it can be interrupted at any time without specific reason and the consent is then signed before the interview is carried out. Signed consent is saved in study folder and a copy is submitted to the participant.

Sound recordings will be made during the interviews and transcribed afterwards. The transcribed interviews will be provided with information on time, place and a serial number for informants and researchers. No personal data is collected together with the interviews.

Archiving of interview data for the qualitative part takes place on digital medium according to current security procedures that ensure that only authorized researchers have access to the material. Recorded material will be unidentified and stored for 10 years as digital audio files in our digital archive. Then the material will be destroyed.

ELIGIBILITY:
Inclusion Criteria:

* Doctors diagnosed asthma

Exclusion Criteria:

* Presence of comorbidity with significant impact on symptom control

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Symptom control | By 6 months
  Mean score of Asthma Control Test, e-questionnaire will be sent to participants to fill in.

SECONDARY OUTCOMES:
Exacerbations | Up to 6 months
  Number of exacerbations, E-questionnaire collecting information about number of exacerbations requiring oral corticosteroids or unplanned healthcare visits or missed school/workdays due to asthma
Adherence | Up to 6 months
  Mean score of participants forgetfulness to ta control medication according to Medicine Adherence Report Scale; 1=always, 2=often, 3=sometimes, 4=rarely, 5=never
Lung function | Up to 12 months, singel arm, only patients allocated to the intervention
  Fluctuation in time-serial measurements (forced expiratory volume in one second FEV1 (L)) according to measurements with Asthmatuner, information will be linked to exacerbations, daily- and nocturnal symptoms as well as treatment with bronchodilator

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Healthcare region Tiohundra, Norrtälje
  - Astrid Lindgren Children's Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared on request and approval from ethic committee